CLINICAL TRIAL: NCT00071136
Title: Phase 1/2 Dose-Escalating Study of Biweekly Alimta and Gemcitabine in Patients With Advanced Cancer
Brief Title: Pemetrexed and Gemcitabine in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7221; H3E-US-JMGC
Record Dates: First submitted 2003-10-13; First posted 2003-10-16 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: pemetrexed
Drug: gemcitabine

SUMMARY:
This is a Phase 2 study of pemetrexed and gemcitabine chemotherapy given once every 14 days to patients with advanced stage non-small cell lung cancer. This treatment is for patients that have not received any prior chemotherapy treatment for lung cancer. The primary goal is to find out if the tumor gets smaller or disappears with this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of advanced stage non-small cell lung cancer.
2. Are able to be active at home and/or work.
3. Have not received chemotherapy for this cancer disease.
4. Have good organ function (for example, most blood work is normal).
5. Have completed any prior radiation treatment at least 4 weeks ago.

Exclusion Criteria:

1. Have been treated with an investigational/research drug within the last month.
2. Have cancer that has spread to the brain and is causing symptoms.
3. Have an active infection or other serious medical condition.
4. Have a second cancer in addition to non-small cell lung cancer.
5. Can not stop taking aspirin or other anti-inflammatory agents for 5-8 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-12; Study Completion 2006-08

PRIMARY OUTCOMES:
To find out how often tumors become smaller or disappear in patients with advanced NSCLC treated with gemcitabine followed by pemetrexed once every 14 days. Chemotherapy treatment will be given for up to 12 times or until the cancer disease increases.

SECONDARY OUTCOMES:
To measure the effects of chemotherapy treatment on:
time until the cancer becomes less;time to cancer re-appears or becomes larger;length of time there is no increase in the amount of cancer;length of time patients survive;
To measure the side-effects from this chemotherapy as given once every 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC-GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC-GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC-GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC-GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC-GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas